CLINICAL TRIAL: NCT06095115
Title: A Phase 3 Multicenter, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy and Safety of JNJ-77242113 for the Treatment of Participants With Moderate to Severe Plaque Psoriasis With Randomized Withdrawal and Retreatment
Brief Title: A Study of JNJ-77242113 in Adolescent and Adult Participants With Moderate to Severe Plaque Psoriasis
Acronym: ICONIC-LEAD
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 77242113PSO3001; 77242113PSO3001 (Other: Janssen Research & Development, LLC); 2023-505120-59-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2023-10-18; First posted 2023-10-23 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Plaque Psoriasis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- JNJ-77242113 (Experimental): Adolescent and adult participants will receive JNJ-77242113 from Week 0 through Week 156. At Week 24, adult participants who are psoriasis area and severity index (PASI) 75 or investigator global assessment (IGA) score of 0 or 1 responders (that is, those who achieve an IGA score of 0 or 1 and have >=2-grade improvement from baseline) will be re-randomized either to continue JNJ-77242113 or to placebo (and will be retreated with JNJ-77242113 upon loss of >=50% of their Week 24 PASI improvement). Adult participants identified as both PASI 75 and IGA 0 or 1 score non-responders will continue to receive JNJ-77242113 through Week 52. From Week 52 to Week 156, all adult participants will receive JNJ-77242113. Adolescents will not participate in re-randomization regardless of their PASI score or IGA score at Week 24. Adolescents will continue to receive JNJ-77242113 from Week 0 through Week 156.
  Interventions: Drug: JNJ-77242113
- Placebo (Experimental): Adolescent and adult participants will receive JNJ-77242113 matching placebo from Week 0 to Week 16. Participants will cross-over to receive JNJ-77242113 from Week 16 through Week 156.
  Interventions: Drug: JNJ-77242113; Drug: Placebo

INTERVENTIONS:
Drug: JNJ-77242113 — JNJ-77242113 will be administered orally.
Drug: Placebo — Placebo will be administered orally
  Arms: Placebo

SUMMARY:
The purpose of this study is see how effective is JNJ-77242113 in participants with moderate to severe plaque psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of plaque psoriasis, with or without psoriatic arthritis, for at least 26 weeks prior to the first administration of study intervention
* Total body surface area (BSA) greater than or equal to (>=)10 percent (%) at screening and baseline
* Total psoriasis area and severity index (PASI) >=12 at screening and baseline
* Total investigator global assessment (IGA) >=3 at screening and baseline
* Candidate for phototherapy or systemic treatment for plaque psoriasis
* A female participant of childbearing potential must have a negative highly sensitive serum pregnancy test beta-human chorionic gonadotropin (beta-hCG) at screening and a negative urine pregnancy test at Week 0 prior to administration of study intervention

Exclusion Criteria:

* Nonplaque form of psoriasis (for example, erythrodermic, guttate, or pustular)
* Current drug-induced psoriasis (for example, a new onset of psoriasis or an exacerbation of psoriasis from beta blockers, calcium channel blockers, or lithium)
* A current diagnosis or signs or symptoms of severe, progressive, or uncontrolled renal, liver, cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurologic, hematologic, rheumatologic, psychiatric, or metabolic disturbances
* Known allergies, hypersensitivity, or intolerance to JNJ-77242113 or its excipients
* Major surgical procedures, (for example, requiring general anesthesia) within 8 weeks before screening, or will not have fully recovered from a surgical procedure or has a surgical procedure planned during the time the participant is expected to participate in the study

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 684 (Actual)
Dates: Start 2023-10-12 (Actual); Primary Completion 2024-07-29 (Actual); Study Completion 2027-04-06 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Achieving an Investigator's Global Assessment (IGA) Score of 0 or 1 and Greater Than or Equal to (>= )2-Grade Improvement From Baseline to Week 16 | Baseline to Week 16
  Percentage of participants who achieve an IGA score of 0 or 1 and >=2-grade improvement from baseline to Week 16 will be reported. The IGA documents the investigator's assessment of the participants psoriasis at a given time point. Overall lesions are graded for induration, erythema, and scaling. The participant's psoriasis is assessed as cleared (0), minimal (1), mild (2), moderate (3), or severe (4).
Percentage of Participants Achieving Psoriasis Area and Severity Index (PASI) 90 Response at Week 16 | Baseline to Week 16
  Percentage of participants achieving PASI 90 response (>=90% improvement in PASI from baseline) at Week 16 will be reported. The PASI is a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. In the PASI system, the body is divided into 4 regions: the head, trunk, upper extremities, and lower extremities. Each of these areas is assessed and scored separately for erythema, induration, and scaling, which are each rated on a scale of 0 to 4 and extent of involvement on a scale of 0 to 6. The PASI produces a numeric score that can range from 0 to 72. A higher score indicates more severe disease.

SECONDARY OUTCOMES:
Percentage of Participants Achieving an IGA Score of 0 at Week 16 | Week 16
  Percentage of participants who achieve an IGA score of 0 at Week 16 will be reported. The IGA documents the investigator's assessment of the participants psoriasis at a given time point. Overall lesions are graded for induration, erythema, and scaling. The participant's psoriasis is assessed as cleared (0), minimal (1), mild (2), moderate (3), or severe (4).
Percentage of Participants Achieving PASI 75 Response at Weeks 4 and 16 | Baseline to Weeks 4 and 16
  Percentage of participants achieving PASI 75 response (>=75% improvement in PASI from baseline) at Weeks 4 and 16 will be reported. The PASI is a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. In the PASI system, the body is divided into 4 regions: the head, trunk, upper extremities, and lower extremities. Each of these areas is assessed and scored separately for erythema, induration, and scaling, which are each rated on a scale of 0 to 4 and extent of involvement on a scale of 0 to 6. The PASI produces a numeric score that can range from 0 to 72. A higher score indicates more severe disease.
Percentage of Participants Achieving PASI 90 Response at Week 8 | Baseline to Week 8
  Percentage of participants achieving PASI 90 response (>=90% improvement in PASI from baseline) at Week 8 will be reported. The PASI is a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. In the PASI system, the body is divided into 4 regions: the head, trunk, upper extremities, and lower extremities. Each of these areas is assessed and scored separately for erythema, induration, and scaling, which are each rated on a scale of 0 to 4 and extent of involvement on a scale of 0 to 6. The PASI produces a numeric score that can range from 0 to 72. A higher score indicates more severe disease.
Percentage of Participants Achieving PASI 100 Response at Week 16 | Week 16
  Percentage of participants achieving PASI 100 response (>=100% improvement in PASI) at Week 16 will be reported. The PASI is a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. In the PASI system, the body is divided into 4 regions: the head, trunk, upper extremities, and lower extremities. Each of these areas is assessed and scored separately for erythema, induration, and scaling, which are each rated on a scale of 0 to 4 and extent of involvement on a scale of 0 to 6. The PASI produces a numeric score that can range from 0 to 72. A higher score indicates more severe disease.
Percentage of Participants Achieving Scalp-specific Investigator Global Assessment (ss-IGA) Score of 0 or 1 and >=2 Grade Improvement Baseline to Week 16 | Baseline to Week 16
  Percentage of participants achieving ss-IGA score of 0 or 1 and >=2 grade improvement baseline to Week 16 will be reported. The ss-IGA instrument is used to evaluate the disease severity of scalp psoriasis. The lesions are assessed in terms of the clinical signs of redness, thickness, and scaliness which are scored as: absence of disease (0), very mild disease (1), mild disease (2), moderate disease (3), and severe disease (4).
Percentage of Participants Achieving Psoriasis Symptoms and Signs Diary (PSSD) Symptom Score of 0 at Weeks 8 and 16 | Weeks 8 and 16
  Percentage of participants achieving PSSD symptom score of 0 at Weeks 8 and 16 will be reported. The PSSD includes patient-reported outcome (PRO) questionnaire designed to measure the severity of psoriasis symptoms and signs over the previous 7 days for the assessment of treatment benefit. The PSSD is a self-administered PRO instrument that includes 11 items covering symptoms (itch, pain, stinging, burning, and skin tightness) and patient-observable signs (skin dryness, cracking, scaling, shedding or flaking, redness, and bleeding) using 0 to 10 numerical rating scales for severity. Two sub scores will be derived each ranging from 0 to 100: the psoriasis symptom score and the psoriasis sign score. A higher score indicates more severe disease.
Percentage of Participants Achieving >=4-Point Improvement From Baseline in PSSD Itch Score to Weeks 4 and 16 | Baseline to Weeks 4 and 16
  Percentage of participants achieving >=4-Point improvement from baseline in PSSD itch score to Weeks 4 and 16 will be reported. The PSSD includes PRO questionnaire designed to measure the severity of psoriasis symptoms and signs over the previous 7 days for the assessment of treatment benefit. The PSSD is a self-administered PRO instrument that includes 11 items covering symptoms (itch, pain, stinging, burning, and skin tightness) and patient-observable signs (skin dryness, cracking, scaling, shedding or flaking, redness, and bleeding) using 0 to 10 numerical rating scales for severity. Two sub scores will be derived each ranging from 0 to 100: the psoriasis symptom score and the psoriasis sign score. A higher score indicates more severe disease.
Time to Loss of PASI 75 | Week 24 up to Week 52
  Time to loss of PASI 75 will be reported. Loss of PASI 75 response is defined as <75% improvement in PASI from Week 24 up to Week 52 in an adult participant who had achieved >=75% improvement in PASI from baseline at Week 24. The PASI is a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. In the PASI system, the body is divided into 4 regions: the head, trunk, upper extremities, and lower extremities. Each of these areas was assessed separately for the percentage of the area involved, which translates to a numeric score that ranges from 0 (indicates no involvement) to 6 (90% to 100% involvement), and for erythema, induration, and scaling, which are each rated on a scale of 0 to 4. The PASI produces a numeric score that can range from 0 (no psoriasis) to 72. A higher score indicates more severe disease. A PASI 75 response represents at least a 75% improvement from baseline in the PASI score.
Time to Loss of PASI 90 | Week 24 up to Week 52
  Time to loss of PASI 90 will be reported. Loss of PASI 90 response is defined as <90% improvement in PASI from Week 24 up to Week 52 in an adult participant who had achieved >=90% improvement in PASI from baseline at Week 24. The PASI is a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. In the PASI system, the body is divided into 4 regions: the head, trunk, upper extremities, and lower extremities. Each of these areas was assessed separately for the percentage of the area involved, which translates to a numeric score that ranges from 0 (indicates no involvement) to 6 (90% to 100% involvement), and for erythema, induration, and scaling, which are each rated on a scale of 0 to 4. The PASI produces a numeric score that can range from 0 (no psoriasis) to 72. A higher score indicates more severe disease. A PASI 90 response represents at least a 90% improvement from baseline in the PASI score.
Number of Participants with Treatment-emergent Adverse Events (AEs) | Up to 160 weeks
  An adverse event (AE) is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the intervention under study. Treatment-emergent AEs are defined as AEs with onset or worsening on or after date of first dose of study treatment.
Number of Participants with Treatment-emergent Serious Adverse Events (SAEs) | Up to 160 weeks
  A SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability or incapacity; congenital anomaly. Treatment-emergent SAEs are defined as serious events between administration of study drug and after the last dose that were absent before treatment or that worsen relative to pretreatment state.
Change from Baseline in Body Surface Area (BSA) at Week 16 | Baseline to Week 16
  Change from baseline in BSA to Week 16 will be reported. BSA is a commonly used measure of extent of skin disease. It is defined as the percentage of surface area of the body involved with the condition being assessed (that is, plaque psoriasis).
Change from Baseline in PASI Total Score to Week 16 | Baseline to Week 16
  Change from baseline in PASI total score to Week 16 will be reported. The PASI is a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. In the PASI system, the body is divided into 4 regions: the head, trunk, upper extremities, and lower extremities. Each of these areas is assessed and scored separately for erythema, induration, and scaling, which are each rated on a scale of 0 to 4 and extent of involvement on a scale of 0 to 6. The PASI produces a numeric score that can range from 0 to 72. A higher score indicates more severe disease.
Percent Improvement in PASI Score From Baseline to Week 16 | Baseline to Week 16
  Percent improvement in PASI score from baseline to Week 16 will be reported. The PASI is a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. In the PASI system, the body is divided into 4 regions: the head, trunk, upper extremities, and lower extremities. Each of these areas is assessed and scored separately for erythema, induration, and scaling, which are each rated on a scale of 0 to 4 and extent of involvement on a scale of 0 to 6. The PASI produces a numeric score that can range from 0 to 72. A higher score indicates more severe disease.
Percentage of Participants Achieving a Static Physician's Global Assessment of Genitalia (sPGA-G) Score of 0 or 1 and at Least a 2-grade Improvement in Genital Psoriasis From Baseline to Week 16 | Baseline to Week 16
  Percentage of participants achieving a sPGA-G Score of 0 or 1 and at Least a 2-grade Improvement in genital psoriasis from baseline to Week 16 will be reported. The sPGA-G is a 6-point scale to assess the severity of genital psoriasis at a given time point. The sPGA-G evaluates erythema, plaque elevation, and scale of genital psoriatic lesions. The severity of genital psoriasis is assessed as clear (0), minimal (1), mild (2), moderate (3), severe (4), and very severe (5).
Percentage of Participants Achieving a Physician's Global Assessment of Hands and Feet (hf-PGA) Score of 0 or 1 and at Least a 2-grade Improvement at Week 16 | Week 16
  Percentage of participants achieving a hf-PGA score of 0 or 1 and at least a 2-grade improvement at Week 16 will be reported. The hf-PGA assesses the severity of hand and foot psoriasis using a 5-point scale to score the plaques on the hands and feet as: clear (0), almost clear (1), mild (2), moderate (3), and severe (4).
Percent Change From Baseline in Modified Nail Psoriasis Severity Index (mNAPSI) Score at Week 16 | Baseline to Week 16
  Percent change from baseline in mNAPSI score at Week 16 will be reported. The mNAPSI is an index used for assessing and grading the severity of nail psoriasis. Each of the participant's 10 fingernails are evaluated for 7 features. The first3 features are each scored from 0 to 3 in severity and are (1) onycholysis and oil-drop dyschromia, (2) pitting, and (3) nail plate crumbling. The next 4 features are scored 0 - absent or 1 - present and are (1) leukonychia, (2) splinter hemorrhages, (3) nail bed hyperkeratosis, and (4) red spots in the lunula. The score ranges from 0 to 13 per nail and 0 to 130 for all fingernails.
Percent of Participants Achieving Fingernail Physician's Global Assessment (f-PGA) Score of 0 or 1 at Week 16 | At Week 16
  Percent of participants achieving f-PGA score of 0 or 1 at Week 16 will be reported. The f-PGA is used to evaluate the current status of a participant's fingernail psoriasis on a scale of 0 to 4 (clear [0], minimal [1], mild [2], moderate [3], or severe [4]).
Change From Baseline in PSSD Symptom Score to Week 16 | Baseline to Week 16
  Change from baseline in PSSD symptom score to Week 16 will be reported. The PSSD includes PRO questionnaire designed to measure the severity of psoriasis symptoms and signs over the previous 7 days for the assessment of treatment benefit. The PSSD is a self-administered PRO instrument that includes 11 items covering symptoms (itch, pain, stinging, burning, and skin tightness) and patient-observable signs (skin dryness, cracking, scaling, shedding or flaking, redness, and bleeding) using 0 to 10 numerical rating scales for severity. Two sub scores will be derived each ranging from 0 to 100: the psoriasis symptom score and the psoriasis sign score. A higher score indicates more severe disease.
Change From Baseline in PSSD Sign Score to Week 16 | Baseline to Week 16
  Change from baseline in PSSD sign score to Week 16 will be reported. The PSSD includes PRO questionnaire designed to measure the severity of psoriasis symptoms and signs over the previous 7 days for the assessment of treatment benefit. The PSSD is a self-administered PRO instrument that includes 11 items covering symptoms (itch, pain, stinging, burning, and skin tightness) and patient-observable signs (skin dryness, cracking, scaling, shedding or flaking, redness, and bleeding) using 0 to 10 numerical rating scales for severity. Two sub scores will be derived each ranging from 0 to 100: the psoriasis symptom score and the psoriasis sign score. A higher score indicates more severe disease.
Percentage of Participants Achieving PSSD Sign Score of 0 at Week 16 | Week 16
  Percentage of participants achieving PSSD sign score of 0 at Week 16 will be reported. The PSSD includes PRO questionnaire designed to measure the severity of psoriasis symptoms and signs over the previous 7 days for the assessment of treatment benefit. The PSSD is a self-administered PRO instrument that includes 11 items covering symptoms (itch, pain, stinging, burning, and skin tightness) and patient-observable signs (skin dryness, cracking, scaling, shedding or flaking, redness, and bleeding) using 0 to 10 numerical rating scales for severity. Two sub scores will be derived each ranging from 0 to 100: the psoriasis symptom score and the psoriasis sign score. A higher score indicates more severe disease.
Percentage of Participants Achieving Genital Psoriasis Sexual Frequency Questionnaire (GenPs-SFQ) Item 2 Score of 0 or 1 at Week 16 | Week 16
  Percentage of participants achieving GenPs-SFQ Item 2 score of 0 or 1 at Week 16 will be reported. The GenPs-SFQ is a 2-item participant-reported instrument used to assess the impact of genital psoriasis on the frequency of sexual activity in the last 7 days. Item 1 assesses overall frequency of sexual activity in the last 7 days (none/zero, once, or 2 or more times), and item 2 assesses how frequently genital psoriasis symptoms have limited the frequency of sexual activity in the last 7 days (never [0], rarely [1], sometimes [2], often [3], or always [4]).
Percentage of Participants Achieving Dermatology Life Quality Index (DLQI) Score of 0 or 1 at Week 16 | Week 16
  Percentage of participants achieving DLQI score of 0 or 1 at Week 16 will be reported. The DLQI is a dermatology specific health-related quality of life (HRQoL) instrument designed to assess the impact of the disease on a participant's HRQoL. It is a 10-item questionnaire that assesses HRQoL over the past week and in addition to evaluating overall HRQoL, can be used to assess 6 different aspects that may affect quality of life: symptoms and feelings, daily activities, leisure, work or school performance, personal relationships, and treatment. The total score ranges from 0 to 30 with a higher score indicating greater impact on HRQoL.
Change From Baseline in Total DLQI Score at Week 16 | Baseline to Week 16
  Change from baseline in total DLQI score at Week 16 will be reported. The DLQI is a dermatology specific HRQoL instrument designed to assess the impact of the disease on a participant's HRQoL. It is a 10-item questionnaire that assesses HRQoL over the past week and in addition to evaluating overall HRQoL, can be used to assess 6 different aspects that may affect quality of life: symptoms and feelings, daily activities, leisure, work or school performance, personal relationships, and treatment. The total score ranges from 0 to 30 with a higher score indicating greater impact on HRQoL.
Change from Baseline in Domain Scores of the Patient-reported Outcomes Measurement Information System-29 (PROMIS-29) Score at Week 16 | Baseline to Week 16
  Change from baseline in domain scores of the PROMIS-29 score at Week 16 will be reported. The PROMIS-29 is a 29-item generic HRQoL survey, assessing each of the 7 PROMIS domains(depression, anxiety, physical function, pain interference, fatigue, sleep disturbance, and ability to participate in social roles and activities) with 4 questions for each domain. The questions are ranked on a 5-point Likert scale. There is also a numerical rating scale that ranges from 0 (No pain) to 10 (Worst pain imaginable) for pain intensity. The raw domain scores are converted to standardized T-scores with a mean of 50 and a standard deviation of 10. Higher scores on anxiety, depression, fatigue, sleep disturbance, and pain interference indicate more severe symptoms. Higher scores on physical function and social participation indicate better health outcomes.
Percentage of Participants Achieving Children's Dermatology Life Quality Index (CDLQI) Score of 0 or 1 at Week 16 | Week 16
  Percentage of participants achieving CDLQI score of 0 or 1 at Week 16 will be reported. The CDLQI is an adapted version of the DLQI for the pediatric population and will be utilized in the adolescent population in this study. The adaption and validation of the CDLQI was undertaken by the original developer of the DLQI to ensure it addressed the specific needs of the pediatric population. The CDLQI is a 10-item instrument that has 4 item response options and a recall period of 1 week. Higher scores indicate greater impact on HRQoL. The instrument is designed for use in children is self-explanatory and can be simply handed to the participant who is asked to fill it in with the help of the child's parent or caregiver.
Change From Baseline in CDLQI at Week 16 | Baseline to Week 16
  Change from baseline in CDLQI at Week 16 will be reported. The CDLQI is an adapted version of the DLQI for the pediatric population and will be utilized in the adolescent population in this study. The adaption and validation of the CDLQI was undertaken by the original developer of the DLQI to ensure it addressed the specific needs of the pediatric population. The CDLQI is a 10-item instrument that has 4 item response options and a recall period of 1 week. Higher scores indicate greater impact on HRQoL. The instrument is designed for use in children is self-explanatory and can be simply handed to the participant who is asked to fill it in with the help of the child's parent or caregiver.
Change From Baseline in the Domain Scores of the PROMIS-25 Pediatric Score at Week 16 | Baseline to Week 16
  Change from baseline in the domain scores of the PROMIS-25 pediatric score at Week 16 will be reported. The PROMIS-25 will be utilized in the adolescent population and is a 25-item generic HRQoL survey. Six PROMIS domains (physical function mobility, anxiety, depressive symptoms, fatigue, peer relationships, pain interference) are each assessed with 4 questions. There is also one 11-point rating scale for pain intensity. The instrument is designed for use in ages 8-17 years of age and can be self-administered.
Percentage of Participants Achieving IGA Score of 0 at Week 52 | Week 52
  Percentage of participants achieving IGA score of 0 at Week 52 will be reported. The IGA documents the investigator's assessment of the participants psoriasis at a given time point. Overall lesions are graded for induration, erythema, and scaling. The participant's psoriasis is assessed as cleared (0), minimal (1), mild (2), moderate (3), or severe (4).
Percentage of Participants Achieving PASI 100 Response at Week 52 | Week 52
  Percentage of participants achieving PASI 100 response (100% improvement in PASI) at Week 52 will be reported. The PASI is a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. In the PASI system, the body is divided into 4 regions: the head, trunk, upper extremities, and lower extremities. Each of these areas is assessed and scored separately for erythema, induration, and scaling, which are each rated on a scale of 0 to 4 and extent of involvement on a scale of 0 to 6. The PASI produces a numeric score that can range from 0 to 72. A higher score indicates more severe disease.
Time to Loss of IGA 0 to 1 Response | Week 24 to Week 52
  Time to loss of IGA 0 to 1 response will be reported. The IGA documents the investigator's assessment of the participants psoriasis at a given time point. Overall lesions are graded for induration, erythema, and scaling. The participant's psoriasis is assessed as cleared (0), minimal (1), mild (2), moderate (3), or severe (4).
Percentage of Adolescent Participants Achieving IGA Score of 0 or 1 and >=2 Improvement From Baseline to Week 52 | Baseline to Week 52
  Percentage of adolescent participants achieving IGA score of 0 or 1 and IGA score >=2 from baseline to Week 52 will be reported. The IGA documents the investigator's assessment of the participants psoriasis at a given time point. Overall lesions are graded for induration, erythema, and scaling. The participant's psoriasis is assessed as cleared (0), minimal (1), mild (2), moderate (3), or severe (4).
Percentage of Adolescent Participants Achieving PASI 75 Response at Week 52 | Baseline to Week 52
  Percentage of adolescent participants achieving PASI 75 response (>=75% improvement in PASI from baseline) at Week 52 will be reported. The PASI is a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. In the PASI system, the body is divided into 4 regions: the head, trunk, upper extremities, and lower extremities. Each of these areas is assessed and scored separately for erythema, induration, and scaling, which are each rated on a scale of 0 to 4 and extent of involvement on a scale of 0 to 6. The PASI produces a numeric score that can range from 0 to 72. A higher score indicates more severe disease.
Percentage of Adolescent Participants Achieving PASI 90 Response at Week 52 | Baseline to Week 52
  Percentage of adolescent participants achieving PASI 90 response (>=90% improvement in PASI from baseline) at Week 52 will be reported. The PASI is a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. In the PASI system, the body is divided into 4 regions: the head, trunk, upper extremities, and lower extremities. Each of these areas is assessed and scored separately for erythema, induration, and scaling, which are each rated on a scale of 0 to 4 and extent of involvement on a scale of 0 to 6. The PASI produces a numeric score that can range from 0 to 72. A higher score indicates more severe disease.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (170):
- United States (46):
  - Medical Dermatology Specialists, Phoenix, Arizona
  - Johnson Dermatology, Fort Smith, Arkansas
  - First OC Dermatology, Fountain Valley, California
  - Center for Dermatology Clinical Research, Fremont, California
  - Integrative Skin Science and Research, Sacramento, California
  - Rady Childrens Hospital San Diego, San Diego, California
  - Southern California Dermatology, Santa Ana, California
  - Clinical Science Institute, Santa Monica, California
  - Bioclinical Research Alliance Inc., Miami, Florida
  - Ziaderm Research LLC, North Miami Beach, Florida
  - Forcare Clinical Research Inc, Tampa, Florida
  - Skin Care Physicians of Georgia, Macon, Georgia
  - Arlington Dermatology, Rolling Meadows, Illinois
  - Northshore Medical Group, Skokie, Illinois
  - Dundee Dermatology, West Dundee, Illinois
  - Dawes Fretzin Clinical Research Group LLC, Indianapolis, Indiana
  - Indiana Clinical Trial Center, Plainfield, Indiana
  - Qualmedica Research, Owensboro, Kentucky
  - Dermatology and Advanced Aesthetics, Lake Charles, Louisiana
  - Allcutis Research, Beverly, Massachusetts
  - Michigan Center of Medical Research, Clarkston, Michigan
  - Minnesota Clinical Study Center, New Brighton, Minnesota
  - Skin Specialists, Omaha, Nebraska
  - Allcutis Research, Portsmouth, New Hampshire
  - Schweiger Dermatology Group, East Windsor, New Jersey
  - Icahn School of Medicine at Mt. Sinai, New York, New York
  - Wilmington Dermatology Center, Wilmington, North Carolina
  - Oakview Dermatology, Athens, Ohio
  - Optima Research, Boardman, Ohio
  - Dermatologists of Central States LLC, Fairborn, Ohio
  - Central Sooner Research, Oklahoma City, Oklahoma
  - Oregon Medical Research Center, Portland, Oregon
  - Oregon Dermatology and Research Center, Portland, Oregon
  - The Pennsylvania Centre for Dermatology, LLC, Exton, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Health Concepts, Rapid City, South Dakota
  - Arlington Research Center, Inc., Arlington, Texas
  - The University of Texas Health Science Center at Houston, Bellaire, Texas
  - Center for Clinical Studies, Houston, Texas
  - Texas Dermatology and Laser Specialists, San Antonio, Texas
  - Center for Clinical Studies, Webster, Texas
  - Springville Dermatology CCT Research, Springville, Utah
  - Virginia Dermatology Skin Cancer Center Pllc, Norfolk, Virginia
  - Frontier Derm Partners CRO, LLC, Mill Creek, Washington
  - Premier Clinical Research, Spokane, Washington
- Argentina (7):
  - ARCIS Salud SRL Aprillus asistencia e investigacion, Buenos Aires
  - Centro Privado de Medicina Familiar, Buenos Aires
  - Derma Internacional S A, Buenos Aires
  - Psoriahue, CABA
  - Centro de Investigaciones Medicas Mar Del Plata, Mar del Plata
  - Instituto De Especialidades De La Salud SRL, Rosario
  - MR Medicina Reumatologica, San Fernando
- Australia (6):
  - Dr Rodney Sinclair Pty Ltd, East Melbourne
  - The Alfred Hospital, Melbourne
  - Kingsway Dermatology & Aesthetics, Miranda
  - ISHI dermatology, Mitcham
  - Royal Melbourne Hospital, Parkville
  - Veracity Clinical Research, Woolloongabba
- Canada (11):
  - Dermatology Research Institute Inc, Calgary, Alberta
  - Rejuvenation Dermatology Clinic Edmonton Downtown, Edmonton, Alberta
  - Dr. Chih ho Hong Medical, Surrey, British Columbia
  - Mediprobe Research Inc., London, Ontario
  - Dr Wei Jing Loo Medicine Professional Corporation, London, Ontario
  - Ryan Clinical Research Inc, Newmarket, Ontario
  - Canadian Dermatology Center, Toronto, Ontario
  - Toronto Research Centre, Toronto, Ontario
  - FACET Dermatology, Toronto, Ontario
  - XLR8 Medical Research, Windsor, Ontario
  - Innovaderm Research Inc., Montreal, Quebec
- China (15):
  - China Japan Friendship Hospital, Beijing
  - Beijing Friendship Hospital Capital Medical University, Beijing
  - Peking University Third Hospital, Beijing
  - The Affiliated Hospital of Bengbu Medical College, Bengbu
  - Hosp. of Chengde Medical University, Chengde
  - Chengdu Second People's Hospital, Chengdu
  - The First Hospital of Jiaxing, Jiaxing
  - Qilu Hospital of Shandong University, Jinan
  - Dermatology Hospital of Jiangxi Province, Nanchang
  - Nanyang First People's Hospital, Nanyang
  - Shanghai skin disease hospital, Shanghai
  - Northeast International Hospital, Shenyang
  - Union Hospital Tongji Medical College of Huazhong University of Science and Technology, Wuhan
  - The Second Affiliated Hospital of Xi'an Jiaotong University, Xi'an
  - Affiliated Hospital of Jiangsu University, Zhenjiang
- France (2):
  - Hopital Prive d'Antony, Antony
  - Centre Hospitalier Victor Dupouy, Argenteuil
- Germany (17):
  - Fachklinik Bad Bentheim, Bad Bentheim
  - Charite - Campus Mitte, Berlin
  - Universitatsklinikum Bonn, Bonn
  - Klinische Forschung Dresden GmbH, Dresden
  - Hautzentrum Dulmen, Dülmen
  - Privatpraxis Dr. Hilton & Partner, Düsseldorf
  - Universitaetsklinikum Frankfurt, Frankfurt am Main
  - Universitaetsklinikum Freiburg, Freiburg im Breisgau
  - Derma-Study-Center Friedrichshafen GmbH, Friedrichshafen
  - Universitaetsklinikum Heidelberg, Heidelberg
  - Hautarztpraxis, Mahlow
  - Universitaetsklinikum Muenster, Münster
  - Klinikum Oldenburg, Oldenburg
  - Hautarztpraxis Mortazawi, Remscheid
  - Universitaetsklinik Tuebingen, Tübingen
  - Hautarztpraxis, Witten
  - CentroDerm GmbH, Wuppertal
- Hungary (8):
  - Pecsi Tudomanyegyetem, Borgyogyaszati Klinika
  - Obudai Egeszsegugyi Centrum Kft, Budapest
  - Derma-B Kft, Debrecen
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
  - Somogy Varmegyei Kaposi Mor Oktato Korhaz, Kaposvár
  - SZTE AOK Szent-Gyorgyi Albert Klinikai Kozpont, Borgyogyaszati és Allergologiai Klinika, Szeged
  - Allergo-Derm Bakos Kft., Szolnok
  - Medmare Egeszsegugyi Es Szolgaltato Bt., Veszprém
- Italy (4):
  - Azienda Di Rilievo Nazionale E Di Alta Specializzazione, Palermo
  - Azienda Ospedaliero Universitaria di Parma, Parma
  - Policlinico Tor Vergata, Roma
  - Istituto Clinico Humanitas, Rozzano
- Japan (8):
  - Teikyo University Hospital, Itabashi Ku
  - Hospital of the University of Occupational and Enviromental Health, Kitakyushu-shi
  - Mito Kyodo General Hospital, Mito
  - Nagoya City University Hospital, Nagoya
  - Kindai University Hospital, Osaka Sayama Shi
  - Tohoku University Hospital, Sendai
  - Tokyo Medical University Hospital, Shinjuku
  - Mie University Hospital, Tsu
- Poland (16):
  - Osteo-Medic s.c A. Racewicz, J Supronik, Bialystok
  - Specderm Poznanska sp j, Bialystok
  - Centrum Kliniczno Badawcze J Brzezicki B Gornikiewicz Brzezicka Lekarze Spolka Partnerska, Elblag
  - Centrum Medyczne dr Rajzer Sp z o o, Krakow
  - Specjalistyczny gabinet dermatologiczny Aplikacyjno Badawczy Marek Brzewski Pawel Brzewski Spolka Cywilna, Krakow
  - Centrum Medyczne Promed, Krakow
  - Dermed Centrum Medyczne Sp z o o, Lodz
  - Centrum Terapii Wspolczesnej J M Jasnorzewska Spolka Komandytowo Akcyjna, Lodz
  - Dermodent Centrum Medyczne Aldona Czajkowska Rafal Czajkowski S C, Osielsko
  - SOLUMED Centrum Medyczne, Poznan
  - Clinical Research Center sp z o o MEDIC R s k, Poznan
  - Dorota Bystrzanowska High-Med. Przychodnia Specjalistyczna, Warsaw
  - Klinika Ambroziak Dermatologia, Warsaw
  - DERMMEDICA Sp.z o.o., Wroclaw
  - Wro Medica, Wroclaw
  - Centrum Medyczne Oporow, Wroclaw
- South Korea (5):
  - Korea University Ansan Hospital, Ansan-si
  - Chosun university hospital, Gwangju
  - CHA Bundang Medical Center, CHA University, Gyeonggi-do
  - Hallym University Sacred Heart Hospital, Gyeonggi-do
  - Asan Medical Center, Seoul
- Spain (11):
  - Hosp. Univ. Fundacion Alcorcon, Alcorcón
  - Hosp. Gral. Univ. Dr. Balmis, Alicante
  - Hosp Clinic de Barcelona, Barcelona
  - Hosp. de La Santa Creu I Sant Pau, Barcelona
  - Hosp. Univ. de Basurto, Bilbao
  - Grupo Dermatologico Y Estetico Pedro Jaen, Madrid
  - Hosp. Gral. Univ. Gregorio Maranon, Madrid
  - Hosp. Univ. Son Espases, Palma de Mallorca
  - Hosp. Clinico Univ. de Santiago, Santiago de Compostela
  - Hosp. Virgen Macarena, Seville
  - Hosp. de Manises, Valencia
- Taiwan (6):
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - National Taiwan University Hospital, Taipei
  - Mackay Memorial Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - National Taiwan University Hospital Hsin Chu Branch, Taoyuan District
  - Linkou Chang Gung Memorial Hospital, Taoyuan District
- Turkey (Türkiye) (4):
  - Hacettepe University Medical Faculty, Ankara
  - Gazi University Medical Faculty, Ankara
  - Erciyes University Medical Faculty, Kayseri
  - Ondokuz Mayis University, Samsun
- United Kingdom (4):
  - London North West University Healthcare NHS Trust, Harrow
  - Guys and St Thomas NHS Foundation Trust, London
  - Royal Berkshire Hospital, Reading
  - Salford Royal Hospital, Salford

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

REFERENCES:
- [Derived] Bissonnette R, Soung J, Hebert AA, Pink AE, Pinter A, Moore AY, Shi Y, Wang WH, Toth DP, Miller-Kassamali M, Cafone J, Jiang J, Li S, DeKlotz CMC, Nunes F, Lebwohl MG. Oral Icotrokinra for Plaque Psoriasis in Adults and Adolescents. N Engl J Med. 2025 Nov 6;393(18):1784-1795. doi: 10.1056/NEJMoa2504187. PMID 41191940